CLINICAL TRIAL: NCT04626999
Title: Effect of Knee Instability Due To Rupture Of Anterior Cruciate Ligament On Cartilage Damage Related To Types of Reconstruction Therapy: In Biomechanic, Biomolecular and Radiological Aspects
Brief Title: Single and Double Bundle ACL Reconstructions, in Term of Cartilage Damage Due to Remaining Instability After Surgery.
Acronym: ACL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ismail Hadisoebroto Dilogo, Professor in Faculty of Medicine, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISMBNNCARTRECON
Record Dates: First submitted 2020-10-22; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Anterior Cruciate Ligament Rupture; Knee Instability; Cartilage Damage
Keywords: knee instability; anterior cruciate ligament rupture; cartilage damage; Single Bundle ACL Reconstruction; Double Bundle ACL Reconstruction; COMP (Cartilage Oligomeric Matrix Protein); MRI T2 Mapping
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Pseudoachondroplasia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Synovial fluid COMP (Active Comparator): Knee joint fluid is aspirated for ELISA COMP examination
  Interventions: Procedure: Single Bundle ACL Reconstruction; Procedure: Double Bundle ACL Reconstruction
- MRI T2 Mapping (Active Comparator): Affected knee is subjected to an MRI T2 mapping examination to see the condition of cartilage
  Interventions: Procedure: Single Bundle ACL Reconstruction; Procedure: Double Bundle ACL Reconstruction
- Instability Examination (Active Comparator): Lachmant Test, Pivot shift test and Rolimeter Measurement
  Interventions: Procedure: Single Bundle ACL Reconstruction; Procedure: Double Bundle ACL Reconstruction

INTERVENTIONS:
Procedure: Single Bundle ACL Reconstruction — Arthroscopy Single Bundle ACL Reconstruction is a procedure to reconstruct the ACL using one bundle.
  The procedure uses Hamstring (Gracillis muscle and Semitendinosus muscle) as a graft.
Procedure: Double Bundle ACL Reconstruction — Arthroscopy Double Bundle ACL Reconstruction is a procedure to reconstruct the ACL using Two bundles (Double bundle).
  The procedure uses Gracillis tendon as a Posterolateral bundle graft and Semitendinosus tendon as an Anteromedial bundle graft.

SUMMARY:
The prevalence of ACL (Anterior Cruciate Ligament) ruptures is relatively high, primarily due to sports and military training injuries. With the advancements of ACL reconstruction therapies, there exist two ways to reconstruct ACL: single-bundle ACL reconstruction (SBACLR) and double-bundle ACL reconstruction (DBACLR). Previous research studies claimed that DBACLR techniques are superior to that of SBACLR, while others stated no notable differences between the two. The variables assessed in previous studies are findings related to the clinical instabilities of the knees (both subjective nor objectives views) and standard radiology examination, such as Xray or MRI. Knee instabilities are the primary goal of ACL reconstructions. Hence this study focuses on finding the dissimilarities between the two previously mentioned techniques by observing the early consequences (subclinically) of knee instabilities towards cartilage damage. The dissimilarities assessments utilize biomolecular tests (ELISA) of cartilage oligomeric matrix protein (COMP) on synovial joint fluid of the knee and knee joint cartilage examination using MRI T2 mapping. Furthermore, there will be a stability (biomechanical) check of the knee joint in the form of a Lachman test, a pivot shift test, and a Rolimeter.

This study requires around 47-52 subjects divided into two operation techniques of SBACLR and DBACLR. To evaluate the results from COMP, MRI T2 mapping, Lachman test, pivot shift test, and Rolimeter, this study is divided into three timeframes: before an operation, three months after post-operation, and six months post-operations. The differences between the test variables are then used as an indicator to assess the cartilage conditions from two operation techniques: SBACLR and DBACLR. Subsequently, the study also examines the possible correlation of each of the resulting variables.

DETAILED DESCRIPTION:
This study utilizes a single-blind randomized clinical trial to evaluate whether the DBACL reconstruction surgery is more suitable than SBACL reconstruction in the subclinical aspect of cartilage damage through a biomolecular examination from the synovial joint fluid COMP and MRI T2 mapping.

This study's estimated time is between two to three years ranging from January 2018 until the end of June 2021.

The samples are randomly divided into two groups: the SBACLR group and the DBACLR group. The sample size for each group was 26 subjects. For the subjects, the accepted inclusion criteria were male, age 18-40 years, total primary AC rupture, injury time 1-12 months, willingness to attend the study, and signed informed consent.

Exclusion criteria include subjects having other ligament injuries in the knee, history of rheumatoid arthritis, severe osteoarthritis Kellgren-Lawrence grading> 2, Body Mass Index (BMI) ≥ 25, fracture around the knee joint or osteochondral avulsion, history of injury with either or both semitendinosus or gracilis muscle, patellofemoral instability, contraindication of anesthesia, and partial ACL rupture.

Drop Out criteria includes: subjects not returning to control, undergoing treatment outside the program, not complying with study protocols, re-injury to the studied knee causing ligament, meniscus or cartilage injury, and postoperative knee infection.

Prospective subjects have been diagnosed with the total loss of ACL and meet the research criteria are explained about the aims and objectives of the study and sign a consent form to participate in the study.

Each subject was assigned to one of the study groups through a simple randomization method: the SBACL reconstruction surgery action group or the DBACL reconstruction surgery action group.

All subjects were examined the Lachman test, pivot test, Rolimeter measurement, MRI T2 mapping, and knee joint fluid for ELISA examination of sfCOMP (synovial fluid COMP) at the time before surgery, the third month, and the sixth month postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 18-40 years
* Total primary ACL rupture
* Injury time 1-12 months
* Willingness to attend the study
* Signed informed consent.

Exclusion Criteria:

* Subjects having other ligament injuries in the knee
* History of rheumatoid arthritis
* Severe osteoarthritis Kellgren-Lawrence grading> 2
* Body Mass Index (BMI) ≥ 25
* Fracture around the knee joint or osteochondral avulsion
* History of injury with either or both semitendinosus or gracilis muscle, patellofemoral instability, contraindication of anesthesia, and partial ACL rupture.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Changes of Synovial fluid Cartilage Oligomeric Matrix Protein (sfCOMP) Concentration from Baseline to 3 months and 6 months | 0,3,6 months
  Sample will be taken from Synovial fluid and and send to laboratory for checking the concentration (ng/mL) of COMP using ELISA (enzyme-linked immunosorbent assay) kits.
Changes of MRI T2 Mapping colour from Baseline to 3 months and 6 months | 0,3,6 months
  The cartilage of the affected knee will be checked using MRI T2 Mapping and the resulting color will be quantitatively assessed in seconds.
Changes of Lachman test score from baseline to 3 months and 6 months | 0,3,6 months
  Anterior instability on the affected knee will be checked using the Lachman test and the score is recorded in millimeter (mm).
Changes of Pivot shift test score from baseline to 3 months and 6 months | 0,3,6 months
  Rotatory instability on the affected knee will be checked using the Pivot shift test and the score is recorded in +1, +2, +3.
Changes of Rolimeter measurement score from baseline to 3 months and 6 months | 0,3,6 months
  Anterior instability on the affected knee will be checked using the Rolimeter tools and the measurement is recorded in millimeter (mm).

CONTACTS AND LOCATIONS:
Overall Officials: Bobby N Nelwan, MD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Fakultas Kedokteran Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia